CLINICAL TRIAL: NCT00239564
Title: An Open-Label Study to Assess the Pharmacokinetics and Pharmacodynamics of IPX054 in Subjects With Parkinson's Disease
Brief Title: Pharmacokinetics and Pharmacodynamics of IPX054 in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPX054-B04-06
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2017-01

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: IPX054; Parkinson disease; Levodopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: carbidopa and levodopa (Experimental): Subjects receive IPX054 100 mg, IPX054 150 mg, IPX054 200 mg, IPX054 250 mg, or IPX054 300 mg to achieve optimum dosage and dosing frequency as directed by the Investigator for 5 weeks.
  Interventions: Drug: IPX054 100 mg; Drug: IPX054 150 mg; Drug: IPX054 200 mg; Drug: IPX054 250 mg; Drug: IPX054 300 mg

INTERVENTIONS:
Drug: IPX054 100 mg — IPX054 containing 25 mg carbidopa and 100 mg levodopa
  Other Names: CD-LD ER 100 mg
Drug: IPX054 150 mg — IPX054 containing 37.5 mg carbidopa and 150 mg levodopa
  Other Names: CD-LD ER 150 mg
Drug: IPX054 200 mg — CD-LD CR containing 50 mg carbidopa and 200 mg levodopa
  Other Names: CD-LD ER 200 mg
Drug: IPX054 250 mg — CD-LD CR containing 62.5 mg carbidopa and 250 mg levodopa
  Other Names: CD-LD ER 250 mg
Drug: IPX054 300 mg — CD-LD CR containing 75 mg carbidopa and 300 mg levodopa
  Other Names: CD-LD ER 300 mg

SUMMARY:
The objective is to compare the pharmacokinetics and pharmacodynamics of IPX054 and carbidopa-levodopa immediate-release tablets in subjects with idiopathic Parkinson's disease who are currently being treated with a stable regimen of carbidopa-levodopa immediate-release tablets.

DETAILED DESCRIPTION:
IPX054 contains two different drugs called levodopa and carbidopa in one tablet.

* levodopa turns into a material called 'dopamine' in your brain. The dopamine helps to improve the symptoms of your Parkinson's disease.
* carbidopa belongs to a group of medicines called 'aromatic amino acid decarboxylase inhibitors'. It helps levodopa work more effectively by slowing the speed at which levodopa is broken down in your body.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease
* Currently being treated with a stable dosage regimen of immediate-release carbidopa-levodopa for at least 3 months.
* Must experience at least 3 episodes of "wearing OFF" symptoms and an average of at least 2 hours of "OFF" time per day.

Exclusion Criteria:

* Diagnosed with atypical parkinsonism
* Prior surgical interventions for Parkinson's disease
* Glaucoma
* Undiagnosed skin lesion or history of melanoma
* Epilepsy or history of seizures

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Parkinsonian disability at Visits 1 and 5 | 36 Days

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (2):
- United States (2):
  - Site 101, Sunnyvale, California
  - Site 102, Lawrence, Kansas

IPD SHARING:
Plan to Share IPD: No